CLINICAL TRIAL: NCT01058096
Title: A Double-Blind, Placebo-Controlled, Evaluation of the Safety and Efficacy of Cariprazine in Patients With Acute Mania Associated With Bipolar I Disorder
Brief Title: Safety and Efficacy of Cariprazine for Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-32
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder; Mania
Keywords: Acute Mania; Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cariprazine (Experimental): Cariprazine 3 mg - 12 mg capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Placebo dose-matching cariprazine capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine.
  Arms: Cariprazine
Drug: Placebo — Patients who meet eligibility criteria will be administered a once daily oral dose of placebo.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of cariprazine monotherapy versus placebo for the treatment of acute manic or mixed episodes associated with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed consent prior to any study specific procedures
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder, as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID) manic or mixed type with or without psychotic symptoms
* Voluntarily hospitalized for current manic episode
* Patients with normal physical examination, laboratory, vital signs,and/ or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of an axis I disorder other than bipolar I disorder that was the primary focus of treatment within the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Diaz, MD, Study Director — Forest Laboratories
Locations (28):
- United States (10):
  - Forest Investigative Site 004, Long Beach, California
  - Forest Investigative Site 005, Riverside, California
  - Forest Investigative Site 007, San Diego, California
  - Forest Investigative Site 009, Chicago, Illinois
  - Forest Investigative Site 006, Lake Charles, Louisiana
  - Forest Investigative Site 001, Flowood, Mississippi
  - Forest Investigative Site 003, Creve Couer, Missouri
  - Forest Investigative Site 008, Cleveland, Ohio
  - Forest Investigative Site 010, Oklahoma City, Oklahoma
  - Forest Investigative Site 002, Houston, Texas
- India (18):
  - Forest Investigative Site 106, Vijayawada, Andhra Pradesh
  - Forest Investigative Site 112, Vizag, Andhra Pradesh
  - Forest Investigator Site 108, Varanasi, Durgakund
  - Forest Investigative Site 103, Ahmedabad, Gujarat
  - Forest Investigative Site 120, Ahmedabad, Gujarat
  - Forest Investigative Site 105, Bangalore, Karnataka
  - Forest Investigative Site 107, Bangalore, Karnataka
  - Forest Investigative Site 118, Mangalore, Karnataka
  - Forest Investigative Site 113, Mangalore, Karnataka
  - Forest Investigative Site 115, Manipal, Karnataka
  - Forest Investigative Site 114, Mysore, Karnataka
  - Forest Investigative Site 101, Aurangabad, Maharashtra
  - Forest Investigative Site 110, Nashik, Maharashtra
  - Forest Investigative Site 111, Pune, Maharashtra
  - Forest Investigative Site 104, Pune, Maharashtra
  - Forest Investigative Site 121, Chennai, Tamil Nadu
  - Forest Investigative Site 109, Kanpur, Uttar Pradesh
  - Forest Investigative Site 119, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] McIntyre RS, Masand PS, Earley W, Patel M. Cariprazine for the treatment of bipolar mania with mixed features: A post hoc pooled analysis of 3 trials. J Affect Disord. 2019 Oct 1;257:600-606. doi: 10.1016/j.jad.2019.07.020. Epub 2019 Jul 5. PMID 31344528
- [Derived] Earley W, Durgam S, Lu K, Ruth A, Nemeth G, Laszlovszky I, Yatham LN. Clinically relevant response and remission outcomes in cariprazine-treated patients with bipolar I disorder. J Affect Disord. 2018 Jan 15;226:239-244. doi: 10.1016/j.jad.2017.09.040. Epub 2017 Sep 25. PMID 29017067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants from 1 investigational site are not included in the analyses due to Good Clinical Practice (GCP) violations.
Period: Double-blind Treatment Phase
Arm/Group | Placebo | Cariprazine
Started | 154 | 158
Completed | 106 | 108
Not Completed | 48 | 50
Not completed — Adverse Event | 11 | 15
Not completed — Insufficient Therapeutic Response | 16 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal of Consent | 17 | 26
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other Unspecified | 2 | 0
Period: Safety Follow-up
Arm/Group | Placebo | Cariprazine
Started | 133 (Not all participants continued to Safety Follow-up.) | 134
Completed | 129 | 130
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine | Total
Number analyzed (Participants) | 154 | 158 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (11.8) | 35.8 (11.4) | 36.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 53 | 112
  Male | 95 | 105 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 149 | 153 | 302
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 33 | 66
  Black/African American | 29 | 33 | 62
  Asian | 88 | 91 | 179
  American Indian or Alaska Native | 3 | 0 | 3
  Other | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 71.86 (20.27) | 69.55 (20.06) | 70.69 (20.17)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.39 (10.64) | 165.21 (10.68) | 165.79 (10.66)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meter(m)^2] | 25.73 (5.98) | 25.24 (5.98) | 25.48 (5.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score at Week 3
Description: The YMRS is an 11-item scale that assesses manic symptoms based on the participant's perception of his or her condition over the previous 48 hours, as well as the physician's clinical observations during the interview. The 11-items are elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, rate and amount of speech, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. The severity of the abnormality for 7-items are rated on a 5-point scale (0-4) and 4-items on a 9-point scale (0-8). The individual scores are summed for a total possible score of 0 (best) to 60 (worst). A negative change from Baseline indicates improvement. Analysis was a mixed model for repeated measurements (MMRM) observed cases (OC), with treatment group, pooled study center, visit, treatment group-by-visit interaction as factors, baseline value and baseline-by-visit interaction as covariates and an unstructured covariance matrix.
Time Frame: Baseline, Week 3
Population: Intent-to-treat Population included all participants who received at least 1 dose of study drug and who had at least 1 post-baseline YMRS assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine
Number analyzed (Participants) | 152 | 158
score on a scale | -15.3 (0.9) | -19.6 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Least Squares Mean Difference = -4.3, 95% CI 2-sided [-6.7 to -1.9] — cariprazine - placebo

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Total Score at Week 3
Description: The CGI-S measures the investigator's assessment of overall severity of the participant's illness compared with the severity of illness in other patients the physician has observed using a 7-point scale (1=Normal, not ill at all to 7=Among the most extremely ill participants). A negative change from Baseline indicates improvement. Analysis was based on a MMRM using the observed cases (OC) data, with treatment group, pooled study center, visit, treatment group-by-visit interaction as factors, baseline value and baseline-by-visit interaction as covariates and an unstructured covariance matrix.
Time Frame: Baseline, Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine
Number analyzed (Participants) | 152 | 158
score on a scale | -1.3 (0.1) | -1.6 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine; Test type: Superiority or Other; p = 0.0027, MMRM analysis; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1] — cariprazine - placebo

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose (Up to 51 days)
Description: Safety Population included all randomized participants who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Cariprazine
Serious Adverse Events (participants affected / at risk) | 5/154 | 6/158
Other Adverse Events (participants affected / at risk) | 69/154 | 110/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=154) | Cariprazine (N=158)
Mania (Psychiatric disorders) | 1 | 3
Akathisia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Social stay hospitalisation (Social circumstances) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=154) | Cariprazine (N=158)
Dyspepsia (Gastrointestinal disorders) | 7 | 17
Nausea (Gastrointestinal disorders) | 10 | 16
Vomiting (Gastrointestinal disorders) | 7 | 16
Constipation (Gastrointestinal disorders) | 10 | 14
Diarrhoea (Gastrointestinal disorders) | 6 | 11
Abdominal Discomfort (Gastrointestinal disorders) | 6 | 8
Pyrexia (General disorders) | 5 | 9
Akathisia (Nervous system disorders) | 8 | 35
Extrapyramidal Disorder (Nervous system disorders) | 3 | 24
Tremor (Nervous system disorders) | 9 | 19
Headache (Nervous system disorders) | 16 | 18
Dizziness (Nervous system disorders) | 6 | 14
Somnolence (Nervous system disorders) | 2 | 10
Restlessness (Psychiatric disorders) | 1 | 10
Insomnia (Psychiatric disorders) | 8 | 9

LIMITATIONS AND CAVEATS:
All participants from 1 investigative site are excluded due to GCP violations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.